CLINICAL TRIAL: NCT02325011
Title: An Open-Label, Randomized, Single-Dose, Two-Sequence, Two-Treatment, Four-Period, Crossover Study to Evaluate the Effects of Fluconazole on the Pharmacokinetics (PK) of Sativex® in Healthy Subjects With Cannabis Experience.
Brief Title: An Study to Evaluate the Effects of Fluconazole on the Pharmacokinetics (PK) of Sativex® in Healthy Subjects With Cannabis Experience.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GWCP1427; 2014-003105-16 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Healthy Subjects
Keywords: Sativex; GW-1000-02; Nabiximols; Fluconazole; Pharmacokinetics; Drug-drug interaction
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 (Experimental): During each of the four Inpatient Periods (Visit 2 to Visit 5 inclusive), healthy subjects with a history of cannabis use will either receive a single dose of Sativex® alone (Treatment A) or a single-dose of Sativex coadministered with the interaction drug, fluconazole (Treatment B) on a repeated, cross-over basis.
  Subjects will be randomly assigned to one of two treatment sequences. Treatment sequence 1 is as follows;
  * Visit 2 (Treatment A)
  * Visit 3 (Treatment B)
  * Visit 4 (Treatment A)
  * Visit 5 (Treatment B)
  The crossover treatments will be separated by a washout period of at least 10 days, but no more than 12 days, between each Sativex® dose.
  Interventions: Drug: Sativex® (Treatment A); Drug: Sativex® and fluconazole concomitantly (Treatment B)
- Treatment Sequence 2 (Experimental): During each of the four Inpatient Periods (Visit 2 to Visit 5 inclusive), healthy subjects with a history of cannabis use will either receive a single dose of Sativex® alone (Treatment A) or a single-dose of Sativex coadministered with the interaction drug, fluconazole (Treatment B) on a repeated, cross-over basis.
  Subjects will be randomly assigned to one of two treatment sequences. Treatment sequence 2 is as follows;
  * Visit 2 (Treatment B)
  * Visit 3 (Treatment A)
  * Visit 4 (Treatment B)
  * Visit 5 (Treatment A)
  The crossover treatments will be separated by a washout period of at least 10 days, but no more than 12 days, between each Sativex® dose.
  Interventions: Drug: Sativex® (Treatment A); Drug: Sativex® and fluconazole concomitantly (Treatment B)

INTERVENTIONS:
Drug: Sativex® (Treatment A) — Each 100 uL actuation (spray) of Sativex contains 27 mg/mL THC and 25 mg/mL CBD plus peppermint flavouring. The study dosage of 10.8 mg THC and 10 mg CBD is delivered as four sprays to the oral mucosa.
  Other Names: Nabiximols; GW-1000-02; THC/CBD spray
Drug: Sativex® and fluconazole concomitantly (Treatment B) — Each 100 uL actuation (spray) of Sativex contains 27 mg/mL THC and 25 mg/mL CBD plus peppermint flavouring. The study dosage of 10.8 mg THC and 10 mg CBD is delivered as four sprays to the oral mucosa.
  Fluconazole 200 mg twice daily (BID) for two days, will be administered at the following time points relative to the Day 1 Sativex dose: 1 hour pre-dose, and approximately 11, 24, and 36 hours post-dose.
  Other Names: Nabiximols; GW-1000-02; THC/CBD spray

SUMMARY:
The study aims to evaluate the effect of fluconazole on the pharmacokinetic (PK) profile of a single oromucosal dose of Sativex® (i.e. how the body absorbs, distributes, metabolises and excretes the drug) in healthy subjects with a history of cannabis use.

The primary clinical hypothesis is that no drug-drug interaction between Sativex® and fluconazole will be detected as effects on PK parameters of Sativex®, when both are administered to healthy human volunteers who have experience using cannabis.

The study additionally aims to evaluate the safety and tolerability of an oromucosal dose of Sativex® in subjects when given concurrently with fluconazole.

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomized, single-dose, two-sequence, two-treatment, four-period, crossover study to evaluate the effects of fluconazole on the PK of Sativex® in healthy subjects with cannabis experience.

Subjects will be randomly assigned to one of the two treatment sequences. Each sequence has four Inpatient Periods. During each Inpatient Period, a subject will either receive a single dose of Sativex® alone (Treatment A) or a single-dose Sativex® coadministered with the interaction drug, fluconazole (Treatment B). The crossover treatments will be separated by a washout period of at least 10 days, but no more than 12 days, between each Sativex® dose.

Specifically in both Treatments A and B, a single oromucosal dose of Sativex® (10.8 mg THC and 10 mg CBD delivered in four sprays) will be administered in a fasted state on Day 1 within each Inpatient Period. During Treatment B, fluconazole 200 mg twice daily (BID) for two days, will be administered at the following time points relative to the Day 1 Sativex® dose: 1 hour pre-dose, and approximately 11, 24, and 36 hours post-dose.

Subjects will be checking into the clinical research facility on Day 1 for each Inpatient Period. Subjects will be confined to the clinical research facility during each Inpatient Period, remaining in the clinical unit after dosing under observation through the collection of all PK blood samples. Fifteen PK blood samples will be taken per subject during each study period: prior to Sativex® dosing (t=0) and at the following multiple time points after dosing: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours; along with some select samples for fluconazole measurements (Day 1 and 2 pre-fluconazole morning dose, 4 hours and 8 hours post-fluconazole morning dose). Subjects will be discharged from the unit after the 48-hour post-dose PK sample and samples for clinical laboratory tests and vital signs have been taken and the subject is determined to be fit for discharge.

A Safety Follow-Up Visit will be performed 7 (+2) days after last Inpatient period.

The expected duration for study participation (including Screening Visit, Inpatient Periods, and Safety Follow-up Visit) for each individual subject is a maximum of 61 days.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects must fulfill ALL of the following criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy, male or female, between 18 and 45 years of age (inclusive).
3. Previous experience with cannabis; "cannabis experience" is defined as use of cannabis in the past, but not within 12 months prior to entry into the study.
4. Able (in the investigator's opinion) and willing to comply with all study requirements.
5. Willing and able to communicate with the investigator.
6. Vital signs at screening (after five minutes resting measured in the supine position) within the following ranges:

   1. Body temperature between 35.0 to 37.5 °C
   2. Systolic blood pressure, 90 to 150 mmHg*
   3. Diastolic blood pressure, 60 to 90 mmHg*
   4. Pulse rate, 40 to 99 beats per minute*. (*Blood pressure and pulse rate will be taken again in a standing position. After two minutes standing, there shall be no more than a 20 mmHg drop in systolic or 10 mmHg drop in diastolic blood pressure, associated with clinical manifestation of postural hypotension).
7. Body mass index (BMI) between 18-30 kg/m2 (both inclusive) as calculated by the following BMI formula: Weight (kg) ÷ [Height (m)]2
8. Willing for his or her name to be reported to the responsible authorities for participation in this study, as applicable in individual countries.
9. Willing to allow his or her primary care practitioner and consultant to be notified of participation in the study.

Exclusion Criteria:

The subject may not enter the study if ANY of the following apply:

1. Donation or loss of 400 mL or more of blood within eight weeks prior to first dosing (Visit 2) and unwilling to abstain from donation of blood during the study.
2. Significant concomitant illness within the two weeks prior to first dosing (Visit 2).
3. At risk for requiring hospital admission or extended hospital stay during the study or any scheduled elective hospitalization during the planned study duration.
4. Has any surgical or medical condition, significant disease or disorder or any finding on physical examination and/or oral examination which might significantly alter the absorption, distribution, metabolism or excretion of drugs or that, in the opinion of the investigator, may put the subject at risk, influence the result of the study, or the subjects' ability to participate in the study.
5. Clinical evidence of acute or chronic liver disease or liver injury as indicated by clinically significant abnormal liver function tests such as aspartate aminotransferase, alanine aminotransferase, gamma glutamyl-transpeptidase, alkaline phosphatase, (any ≥2.5 upper limit of normal [ULN]) or serum bilirubin (≥1.5 ULN) unless there is another more likely explanation (eg, Gilbert's syndrome).
6. Significant renal disease or significantly impaired renal function with an estimated creatinine clearance below 50 mL/min.
7. Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP, Sativex.
8. Have a history of known hypersensitivity or idiosyncratic reaction to fluconazole, its excipients, or related compounds.
9. Positive result for the presence of hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCAb), or HIV I or II antibodies.
10. Currently using or has used cannabis and/or cannabinoid based medications (eg, Marinol®, Nabilone®, Cannador®) or Acomplia (rimonabant) or taranabant within 12 months prior to first dosing (Visit 2) and is unwilling to abstain for the duration of the study.
11. Currently using or has used an illicit drug or non prescribed use of any prescription drug within 12 months prior to first dosing (Visit 2) and is unwilling to abstain for the duration of the study.
12. Any known or suspected history of a substance abuse/dependence disorder within the 12 months prior to first dosing (Visit 2).
13. Has a positive urine drug (including THC) or alcohol result at screening or on Day -1 of Visit 2.
14. Current heavy alcohol consumption (more than 60 g of pure alcohol per day for men, and more than 40 g of pure alcohol per day for women).
15. Unwilling to abstain from drinking alcohol during this study (for 24 hours prior to, and for the duration of, each study visit).
16. Had any treatment with any known enzyme-altering agents (barbiturates, phenothiazines, cimetidine, etc.) within 30 days prior to first dosing (Visit 2) or during the study.
17. Unwilling to abstain from nicotine products from midnight Day -1 to 48 hours postdose for each Inpatient Period.
18. Unwilling to abstain from grapefruit products for one week prior to and throughout the Inpatient Period.
19. Have had substantial changes in eating habits, per the investigator's opinion, within 30 days prior to screening.
20. Consume more than five caffeinated beverages per day (eg, five cups of tea or coffee or cans of cola) or who are unwilling to abstain from consumption of caffeine-containing food and beverages throughout each Inpatient Period.
21. Any known or suspected history or immediate family history of schizophrenia, or other psychotic illness, history of severe personality disorder or other severe significant psychiatric disorder other than depression associated with underlying condition.
22. Any history of epilepsy as evidenced by one or more seizures in the last 12 months.
23. Significant cardiac disease, or a cardiac disorder that in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction, or has a secondary or tertiary atrioventricular block, or evidence of clinically significant cardiac disease on ECG at screening.
24. Sexually active males whose partner is of childbearing potential who do not agree to practice two highly effective methods of birth control or remain abstinent during the study and for three months after the last dose of IMP. Sexually active females of childbearing potential who do not agree to practice two highly effective methods of birth control or remain abstinent during the study and for three months after the last dose of IMP. If employing birth control, two of the following precautions must be used: established use of oral, transdermal, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system (consideration should be given to the type of device or system being used, as there are higher failure rates quoted for certain types, eg, steel or copper wire); Condoms with spermicidal foam/ gel/ film/ cream/ suppository; the use of a condom should always be supplemented with the use of a spermicide. Male sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). True abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.

    Note: Non-childbearing potential is defined as female subjects who are surgically sterile (ie, have undergone bilateral salpingo-oophorectomy, hysterectomy) and female subjects who have been postmenopausal for at least 12 consecutive months.
25. Pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
26. Received an IMP within 30 days or five times the t½ of the IMP (whichever is greater) prior to the Screening Visit.
27. Travel outside the country of residence planned during the study.
28. Use of any prescription medication or over-the-counter medication within 14 days prior to Screening or during the study.
29. Previously enrolled in this study or another Sativex study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of Δ9 Tetrahydrocannabinol (THC): Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for THC:
  * Mean maximum (peak) plasma concentration of the drug (Cmax)
  * Mean area under the concentration-time curve calculated to the last observable concentration at time t (AUC(0-t))
  * Mean area under the concentration-time curve from time zero to infinity (AUC(0-∞))
Pharmacokinetic parameters of 11-hydroxy-THC (11-OH-THC): Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for 11-OH-THC:
  * Mean Cmax
  * Mean AUC(0-t)
  * Mean AUC(0-∞)
Pharmacokinetic parameters of Cannabidiol (CBD): Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for CBD:
  * Mean Cmax
  * Mean AUC(0-t)
  * Mean AUC(0-∞)
Pharmacokinetic parameters of 7-hydroxy-CBD (7-OH-CBD): Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for 7-OH-CBD:
  * Mean Cmax
  * Mean AUC(0-t)
  * Mean AUC(0-∞)

SECONDARY OUTCOMES:
Pharmacokinetic parameters of THC: t(1/2), tmax and CL/F | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for THC;
  * Mean terminal-phase elimination half-life (t(1/2))
  * Mean time to maximum (peak) plasma concentration (tmax)
  * Mean apparent clearance of drug from plasma (CL/F)
Pharmacokinetic parameters of 11-OH-THC: t(1/2) and tmax | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for 11-OH-THC;
  * Mean t(1/2)
  * Mean tmax
Pharmacokinetic parameters of CBD: t(1/2), tmax and CL/F | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for CBD;
  * Mean t(1/2)
  * Mean tmax
  * Mean CL/F
Pharmacokinetic parameters of 7-OH-CBD: t(1/2) and tmax | Pre-dose (t=0) and up to 48 hours post-dose (for each of the four treatment periods)
  The following are presented for 7-OH-CBD;
  * Mean t(1/2)
  * Mean tmax
The incidence of adverse events as a measure of subject safety | From screening to follow-up (a maximum of 61 days)
  The number of subjects who experienced an adverse event during the study is presented. The time-frame for adverse event reporting was from screening to the follow-up visit.
The number of subjects with a clinically significant change in physical and oral examination results, relative to pre-treatment baseline | From screening to follow-up (a maximum of 61 days)
  The number of subjects with a change in physical and oral examination results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in 12-lead electrocardiogram (ECG) results, relative to pre-treatment baseline | From screening to follow-up (a maximum of 61 days)
  The number of subjects with a change in ECG results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with clinically significant changes in laboratory test parameters, relative to pre-treatment baseline | From screening to follow-up (a maximum of 61 days)
  The number of subjects with clinically significant changes in serum biochemistry, haematology and urinalysis, relative to the pretreatment baseline, is presented.
The number of subjects with a clinically significant change in vital signs, relative to pre-treatment baseline | From screening to follow-up (a maximum of 61 days)
  The number of subjects with a clinically significant change in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate) indicative of an adverse event, relative to the pre-treatment baseline, is presented.
  A clinically significant drop in blood pressure is defined as a 20 mmHg drop in systolic or 10 mmHg drop in diastolic blood pressure associated with a clinical manifestation of postural hypotension after two minutes standing.

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States